CLINICAL TRIAL: NCT04275154
Title: Evaluating Immunological Parameters, Neurocognitive Changes, Activity Levels, and Driving Fitness in Hematological Malignancy Patients Undergoing Chimeric Antigen Receptor (CAR)-T Cell Therapy
Brief Title: Immunological Parameters, Neurocognitive Changes, Activity, & Driving Fitness in Patients Undergoing CAR-T Cell Therapy
Status: Withdrawn | Type: Observational
Why Stopped: Covid-19 did suspend the study for a period, then when trying to re-open the collaborating department had restructured fees which made it impossible to do the study with the limited grant funds available for this project.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0157-19-FB
Record Dates: First submitted 2020-02-14; First posted 2020-02-19 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Hematologic Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We expect that serum inflammatory cytokine protein concentrations will be elevated in patients showing symptoms of high-grade CRS relative to patients showing symptoms of low-grade or no CRS. We expect that CRS grade will be positively associated with changes in concentrations of IL-6, IL-10, IFN-gamma, and TNF-alpha.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CAR-T patients: Relapsed or refractory Diffuse large B-cell lymphoma (DLBCL) or acute lymphoblastic leukemia (ALL) with intent to undergo commercially available CAR-T cell therapy

SUMMARY:
Chimeric antigen receptor (CAR) T-cell therapy is a promising new treatment that re-programs patient immune cells to target and destroy cancer cells. Importantly, CAR T-cell therapy has improved overall response rate and durability in patients with refractory or relapsed diffuse large B-cell lymphoma (DLCBL) and acute lymphoblastic leukemia (ALL).

Toxicities following CAR T-cell therapy remain a major limitation to expanding access to this promising cancer treatment. Biological predictors of CAR-T-related toxicities are currently lacking, and it remains unknown whether CAR-T-related toxicities lead to subsequent impairments in instrumental activities of daily living. The overarching goal of this project aims to link biological predictors of CAR-T-related toxicities to instrumental activities of daily living, such as physical activity and driving performance. The current study proposes to test the hypothesis that CAR T-cell therapy causes changes in immunological and neurological markers that predict changes in physical activity levels and driving performance.

DETAILED DESCRIPTION:
Study specific aims are: (1A) Evaluate changes in serum inflammatory cytokine protein markers in patients receiving CAR T-cell therapy; (1B) Evaluate changes in electroencephalographic and radiologic markers of CAR-T-related toxicities in comparison to neurocognitive function following CAR T-cell therapy; (2A) Assess changes in activity levels using actigraphy/accelerometry to continuously monitor physical activity; and (2B) Assess changes in driving performance using a standardized on-road instrumented vehicle drive.

Patients (n=20) will be recruited into the study if they are diagnosed with relapsed or refractory DLBCL or ALL, and scheduled to undergo commercially-available CAR T-cell therapy.

The following measures will be completed during primary study visits: prior to apheresis (T0) and 8-weeks post CAR-T cell infusion (T6). (1) blood inflammatory proteins; (2) brain wave recordings (or EEG), brain imaging, and neurocognitive assessment; (3) free-living activity levels; and (4) driving performance and safety. EEG will assess neural activity patterns of brain dysfunction; brain imaging will look for brain abnormalities; neurocognitive assessments will evaluate changes in thinking, concentration, and memory. A research-grade activity monitor will be used to assess activity levels. Driving performance and safety will be evaluated using a driving simulator and an on-road vehicle designed to monitor behavior while drivers complete a driving course. Analyses will assess changes between study visits, as well as relationships between immunological, neurological, activity, and driving measures.

ELIGIBILITY:
Inclusion Criteria:

1. R/R DLBCL or R/R ALL diagnosis
2. Scheduled to receive commercial CAR-T cell therapy (Axi-Cel or Tisagenlecleucel)
3. greater than or equal to 19 years of age
4. Legally licensed to drive for at least 5 years
5. Previously drove an average of 50 miles/week or at least 1 hour/week
6. Normal visual acuity (20/40 or better)
7. Fluent in English

Exclusion Criteria:

(1) Cognitive impairment (MMSE score < 21) prior to baseline assessment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Relapsed or refractory DLBCL or ALL with intent to undergo commercially available CAR-T cell therapy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Evaluate the relationship between immunologic markers of CRS and ICANS in hematologic malignancy patients undergoing CAR-T cell therapy | 6 weeks
  Change in serum inflammatory cytokine (IL-2, IL-4, IL-6, IL-10, TNF-alpha IFN-gamma, and IL-17A) concentrations from baseline
Evaluate the relationship between neurologic markers of CRS and ICANS in hematologic malignancy patients undergoing CAR-T cell therapy | 6 weeks
  Change in number of pathological EEG events from baseline
Activity level parameters- daily number of steps | 6 weeks
  Change in daily number of steps from baseline
On-Road Driving Performance | 6 weeks
  Change in number of driving safety errors from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Lunning, DO, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No